CLINICAL TRIAL: NCT00284206
Title: An Open-Label Trial of Long-Acting Injectable Risperidone in the Treatment of Methamphetamine Dependence
Brief Title: A Trial of Long-Acting Injectable Risperidone in the Treatment of Methamphetamine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: Janssen, LP (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIS-NAP-4008
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Methamphetamine Dependence
Keywords: methamphetamine, cognition, outpatient, risperidone

INTERVENTIONS:
Drug: long-acting injectable risperidone

SUMMARY:
Objective of the Project.

-Methamphetamine (MA) use is growing to epidemic proportions and existing treatments for MA dependence demonstrate sub-optimal efficacy. Research implicates heavy use of MA as at least a contributing agent to a variety of neuropsychiatric impairments including psychosis, mood disturbance, anxiety, cognitive deficits, and motor dysfunction. Initial study by this investigator suggests that agents like risperidone may also be beneficial to MA dependent individuals by decreasing MA use and improving cognitive function in early abstinence. Long-acting injectable risperidone may prove more efficacious given its receptor binding characteristics and potential to increase medication adherence. The study objective is to determine the safety and efficacy of treating MA dependence and the associated cognitive and psychiatric symptomatology with long-acting injectable risperidone.

DETAILED DESCRIPTION:
Objective of the Project.

-Methamphetamine (MA) use is growing to epidemic proportions and existing treatments for MA dependence demonstrate sub-optimal efficacy. Research implicates heavy use of MA as at least a contributing agent to a variety of neuropsychiatric impairments including psychosis, mood disturbance, anxiety, cognitive deficits, and motor dysfunction. Initial study by this investigator suggests that agents like risperidone may also be beneficial to MA dependent individuals by decreasing MA use and improving cognitive function in early abstinence. Long-acting injectable risperidone may prove more efficacious given its receptor binding characteristics and potential to increase medication adherence. The study objective is to determine the safety and efficacy of treating MA dependence and the associated cognitive and psychiatric symptomatology with long-acting injectable risperidone.

Research Plan.

-This is an open-label trial of long-acting injectable risperidone administered 25mg every 2-weeks for the treatment of methamphetamine (MA) dependence. Participation will last approximately 14 weeks. A total of 20 subjects (veterans and non-veterans) aged 18 to 65 years old who meet DSM-IV criteria for current MA dependence, have a stable address or alternative contact, and expect to be in the Puget Sound area for the length of the study will be enrolled at the Seattle and American Lake Divisions of the VA PSHCS. Exclusionary criteria include: 1) known sensitivity or allergy to risperidone; 2) current treatment with an antipsychotic agent, a mood stabilizer, or CYP 2D6 inhibitor; (3) transaminase levels >5X ULN; (4) albumin levels <3.5g/dl; (5) random serum glucose levels >200mg/dl; (6) diabetes mellitus or history of myocardial infarction; (7) baseline Brief Psychiatric Rating Scale score >72; (8) presence of tardive dyskinesia; (9) Barnes Akathisia Rating Scale global item score >2; (10) Simpson-Angus Scale total score > 0.3; (11) involvement with the legal system that could compromise study participation; (12) pregnancy or nursing; (13) receiving current mental health treatment.

Methodology

-Potential subjects will complete a screening, including medical history and physical, laboratory, EKG, assessment of MA and other drug use, psychiatric screening and cognitive testing, to determine eligibility. Eligible subjects will repeat the cognitive testing instruments prior to starting medication. After completing the screening period, subjects who continue to be eligible will receive 7 days of oral risperidone to assess tolerability followed by administration of long-acting injectable risperidone, 25mg. For 3 weeks following the first IM injection, participants will take oral risperidone each night to achieve a therapeutic plasma level of risperidone. During the oral co-administration phase, participants will have medication pill counts during their weekly visit to evaluate adherence and corroborate self-report data. Participants will receive additional 25mg risperidone injections every 14 days (at weeks 2, 4, and 6 after the first injection).

Following the first injection, subjects will return to the study center for weekly visits for 8 weeks. At each study visit, patients will be evaluated for possible adverse events, use of concomitant medications, and use of methamphetamine. Safety labs will be repeated at week 4 and 8. Plasma levels of risperidone and 9-OH-risperidone will be obtained at 3, 6, and 8 weeks. If intolerable adverse events occur, risperidone dosage will be reduced, or, if indicated, risperidone will be discontinued. Psychiatric symptoms and cognitive functioning will be evaluated at Baseline, and 4 and 8 weeks. A follow-up visit will take place at 12 weeks. Subjects will receive behavioral treatment consisting of individual, once weekly, standardized, manual guided, relapse prevention therapy.

Findings, results, or conclusions reached to date.

-None to date.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for methamphetamine (MA) dependence during the past year with current MA use within the 30-days prior to study entry
* Plans to remain in the Puget Sound area for the following 12 weeks
* If female of child bearing potential, agreeable to using an adequate method of birth control
* Age 18-65 years old
* Willing and capable of providing informed consent
* Presence of one or more of the following: stable address, telephone number, or alternative contact person

Exclusion Criteria:

* Known sensitivity or allergy to risperidone
* Current treatment with an antipsychotic agent
* Current treatment with a mood stabilizer
* Current treatment with a CYP 2D6 inhibitor (includes Amiodarone, Bupropion, Celecoxib, Cimetidine, Chlorpromazine, Clomipramine, Fluoxetine, Haloperidol, Methadone, Moclobemide, Paroxetine, Quinidine, Ritonavir, Sertraline, Terbinafine and Thioridazine)
* Presence of tardive dyskinesia
* A global item score >2 on the Barnes Akathisia Rating Scale.
* A total score on the Simpson-Angus Scale > 0.3.
* Albumin level <3.5g/dl.
* Random serum glucose level >200mg/dl.
* Transaminase levels > 5X ULN
* Presence of one or more of the following medical conditions: diabetes mellitus or history of myocardial infarction.
* A total score on the Brief Psychiatric Rating Scale >72.
* Involvement with the legal system that could compromise study participation
* Pregnancy or nursing
* Receiving concurrent mental health treatment in addition to the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Efficacy will be assessed by obtaining weekly self-report measures of MA and other substance use via the timeline follow-back interview corroborated with weekly urine toxicology specimens for substances of abuse including amphetamines.

SECONDARY OUTCOMES:
Secondary efficacy measures include:
changes in neuropsychological performance,
changes in psychiatric symptomatology,
by changes in addiction severity

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Saxon, Principal Investigator — VA Puget Sound Health Care System, and University of Washington Dept. of Psychiatry and Behavioral Sciences
Locations (1):
- VA Puget Sound Health Care System, Addictions Treatment Center, Seattle, Washington, United States